CLINICAL TRIAL: NCT05077800
Title: A Phase II Study of FOLFIRINOX Combined With the Glycogen Synthase Kinase-3 Beta (GSK-3 β) Inhibitor Elraglusib and the Transforming Growth Factor-β (TGF-β) Inhibitor Losartan in Patients With Untreated Metastatic Pancreatic Adenocarcinoma
Brief Title: FOLFIRINOX + Elraglusib + Losartan In Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Colin D. Weekes, M.D., PhD (Other)
Collaborators: Actuate Therapeutics Inc. (Industry); Lustgarten Foundation (Other)
Responsible Party: Sponsor-Investigator, Colin D. Weekes, M.D., PhD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-350
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma Metastatic
Keywords: Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma Metastatic
MeSH Terms: interventions — Losartan; 3-(5-fluorobenzofuran-3-yl)-4-(5-methyl-5H-(1,3)dioxolo(4,5-f)indol-7-yl)-pyrrole-2,5-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Safety Run-In: FOLFIRINOX + Elraglusib + Losartan (Experimental): The study will begin with a Safety Run-In phase to establish the side effects from the study treatment to its safety before beginning the main part of the study, six (6) participants will receive 1-2 cycles (each study cycle is 14 days +/- 3 days) of:
  * FOLFIRINOX
    * 5Fluorouracil portion of FOLFIRINOX on Days 1-3 of each study cycle
    * Irinotecan portion of FOLFIRINOX on Day 1 of each study cycle
    * Oxaliplatin portion of FOLFIRINOX on Day 1 of each study cycle
    * Leucovorin portion of FOLFIRINOX on Day 1 of each study cycle
  The FOLFIRINOX treatment regimen will be given every 14 days +/- 3 days at physician discretion.
  * Elraglusib on days on days 1, 3, 8, and 11 of every 14-day cycle
  * Losartan daily of every 14-day cycle.
  Interventions: Drug: FOLFIRNINOX; Drug: Losartan; Drug: 9-ING-41
- FOLFIRNINOX (Experimental): The study will be conducted in three parts depending on participant disease progression: Complete Therapy, Maintenance Therapy and Complete Therapy Round 2.
  For initial complete therapy, participants will receive FOLFIRINOX as follows (each study cycle is 14 days +/- 3 days, FOLFIRINOX can be given +/- 3 days):
  * 5Fluorouracil portion of FOLFIRINOX on Days 1-3 of each study cycle up to 12 cycles (24 weeks)
  * Irinotecan portion of FOLFIRINOX on Day 1 of each study cycle up to 12 cycles (24 weeks)
  * Oxaliplatin portion of FOLFIRINOX on Day 1 of each study cycle up to 12 cycles (24 weeks)
  * Leucovorin portion of FOLFIRINOX on Day 1 of each study cycle up to 12 cycles (24 weeks)
  For Maintenance therapy, participants will receive FOLFIRINOX as follows:
  * 5Fluorouracil portion of FOLFIRINOX on Days 1-3 of each 14 day study cycle until disease progression For Complete Therapy Round 2, participants will repeat initial complete therapy of FOLFIRINOX until further disease progression
  Interventions: Drug: FOLFIRNINOX
- FOLFIRINOX + Losartan (Experimental): The study will be conducted in three parts depending on participant disease progression: Complete Therapy, Maintenance Therapy and Complete Therapy Round 2.
  For initial complete therapy (each study cycle is 14 days +/- 3 days):
  * FOLFIRINOX (+/- 3 days)
    * 5Fluorouracil portion of FOLFIRINOX on Days 1-3 of each study cycle up to 12 cycles (24 weeks)
    * Irinotecan portion of FOLFIRINOX on Day 1 of each study cycle up to 12 cycles (24 weeks)
    * Oxaliplatin portion of FOLFIRINOX on Day 1 of each study cycle up to 12 cycles (24 weeks)
    * Leucovorin portion of FOLFIRINOX on Day 1 of each study cycle up to 12 cycles (24 weeks)
  * Losartan daily up to 12 cycles (24 weeks)
  For Maintenance therapy:
  * 5Fluorouracil portion of FOLFIRINOX on Days 1-3 of each 14 day study cycle until disease progression
  * Losartan daily until disease progression
  For Complete Therapy Round 2, participants will repeat initial complete therapy of FOLFIRINOX + Losartan until further disease progression
  Interventions: Drug: FOLFIRNINOX; Drug: Losartan
- FOLFIRINOX + Elraglusib (Experimental): The study conducted in 3 parts depending on disease progression: Complete Therapy, Maintenance Therapy and Complete Therapy Round 2
  For initial complete therapy (each study cycle is 14 days +/- 3 days):
  * FOLFIRINOX (+/- 3 days)
    * 5Fluorouracil portion of FOLFIRINOX on Days 1-3 of each study cycle up to 12 cycles (24 weeks)
    * Irinotecan portion of FOLFIRINOX on Day 1 of each study cycle up to 12 cycles (24 weeks)
    * Oxaliplatin portion of FOLFIRINOX on Day 1 of each study cycle up to 12 cycles (24 weeks)
    * Leucovorin portion of FOLFIRINOX on Day 1 of each study cycle up to 12 cycles (24 weeks)
  * Elraglusib on days 1, 3, 8, and 11 of every study cycle up to 12 cycles (24 weeks)
  For Maintenance therapy:
  * 5Fluorouracil portion of FOLFIRINOX on Days 1-3 of each study cycle until disease progression
  * Elraglusib on days 1, 3, 8, and 11 of every study cycle until disease progression For Complete Therapy Round 2, repeat of initial complete therapy until further disease progression
  Interventions: Drug: FOLFIRNINOX; Drug: 9-ING-41
- FOLFIRINOX + Elraglusib + Losartan (Experimental): The study conducted in 3 parts depending on disease progression: Complete Therapy, Maintenance Therapy and Complete Therapy Round 2.
  For initial complete therapy (each study cycle is 14 days +/- 3 days):
  * FOLFIRINOX (+/- 3 days)
    * 5Fluorouracil portion of FOLFIRINOX on Days 1-3 of each study cycle
    * Irinotecan portion of FOLFIRINOX on Day 1 of each study cycle
    * Oxaliplatin portion of FOLFIRINOX on Day 1 of each study cycle
    * Leucovorin portion of FOLFIRINOX on Day 1 of each study cycle
  * Elraglusib on days 1, 3, 8, and 11 of every 14-day cycle
  * Losartan daily
  For Maintenance therapy:
  * 5Fluorouracil portion of FOLFIRINOX on Days 1-3 of each 14 day study cycle until disease progression
  * Elraglusib on days 1, 3, 8, and 11 of every 14-day cycle until disease progression
  * Losartan daily until disease progression
  For Complete Therapy Round 2, participants will repeat initial complete therapy of FOLFIRINOX + Elraglusib + Losartan until further disease progression
  Interventions: Drug: FOLFIRNINOX; Drug: Losartan; Drug: 9-ING-41

INTERVENTIONS:
Drug: FOLFIRNINOX — Combination of 4 different drugs (5-Fluorouracil (5-FU), Oxaliplatin, Irinotecan and Leucovorin) administered by intravenous infusion
Drug: Losartan — Taken Orally
  Other Names: Cozaar
  Arms: FOLFIRINOX + Elraglusib + Losartan; FOLFIRINOX + Losartan; Safety Run-In: FOLFIRINOX + Elraglusib + Losartan
Drug: 9-ING-41 — Administered by intravenous infusion
  Other Names: Elraglusib
  Arms: FOLFIRINOX + Elraglusib; FOLFIRINOX + Elraglusib + Losartan; Safety Run-In: FOLFIRINOX + Elraglusib + Losartan

SUMMARY:
The purpose of this study is to find out if an experimental drug will prevent metastatic pancreatic adenocarcinoma from becoming resistant to standard treatment for the disease.

The names of the study drugs involved in this study are:

* 9-ING-41
* Losartan
* Ferumoxytol
* FOLFIRINOX (made up of 4 different drugs):

  * 5-Fluorouracil (5-FU)
  * Oxaliplatin
  * Irinotecan
  * Leucovorin

DETAILED DESCRIPTION:
This is a multi-institutional, open label, four-arm, non-comparator Phase 2 study of FOLFIRINOX in combination with 9-ING-41 and losartan for the treatment of adult patients with untreated metastatic pancreatic adenocarcinoma (PAC). This research study will begin with a Safety Run-In phase. The Safety Run-In phase will establish the side effects from the study treatment to its safety before beginning the main part of the study. Once that is complete, the main portion of the study will be a Phase II clinical trial.

The U.S. Food and Drug Administration (FDA) has not approved 9-ING-41 as a treatment for pancreatic adenocarcinoma (PAC). The FDA has not approved Losartan for pancreatic adenocarcinoma (PAC), but it has been approved for other uses. The FDA has approved FOLFIRINOX as a treatment option for pancreatic adenocarcinoma (PAC).

This research study involves giving participants an investigational drug called 9- ING-41 with standard anti-cancer drugs. 9-ING-41 stops an enzyme called GSK- 3β from working in cancer cells. Enzymes are proteins that activate and accelerate chemical reactions. The GSK-3β enzyme helps cancer cells to grow and to become resistant to chemotherapy drugs. This study is trying to see if by stopping the activity of GSK-3β using 9-ING-41, it may be possible for standard of care chemotherapy drugs to regain their effectiveness in treating cancers in participants where they have stopped being effective or are effective in only a minority of participants. FOLFIRINOX is a combination of 4 chemotherapy agents that may help shrink pancreatic adenocarcinoma (PAC) tumors. Losartan is a drug that is used to lower blood pressure. In this setting, Losartan has also been demonstrated to suppress TGF-β function in pancreatic adenocarcinoma. Cytokines are molecules that help cells communicate and play a role in immune response. Suppression of TGF-β function is believed to stop the cancer cells from becoming resistant to chemotherapy. This study will evaluate if blocking of GSK-3β activity using 9-ING-41 and blocking of TGF-β function using Losartan can inhibit cancer cell resistance to FOLFIRINOX chemotherapy.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits. Participants will receive treatment during three portions of the study: Complete therapy, Maintenance therapy and Transition to complete therapy. After treatment, participants will be followed for up to 5 years.

It is expected that up to 70 people will take part in this research study.

Actuate Therapeutics, a pharmaceutical company, is supporting this research study by providing the study drug 9-ING-41.

The Lustgarten Foundation is providing funding support for this study through a research grant.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic pancreatic adenocarcinoma without prior therapy for pancreatic adenocarcinoma.
* Participants must have measurable disease as defined by RECIST 1.1
* Age ≥18 years.
* ECOG performance status ≤1 (Karnofsky ≥ 70%, see Appendix A).
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN) if no biliary stenting has been done OR 2.0 x ULN if patient is status post biliary stenting or two downward trending values.
  * AST(SGOT)/ALT(SGPT) < 5 x institutional ULN.
  * Creatinine ≤ 1.5 mg/dL OR .
  * Creatinine clearance ≥ 30 mL/min (as estimated by Cockcroft Gault Equation)

    (140 - age [yrs]) (body wt [kg]) Creatinine clearance for males = ------------ (72) (serum creatinine [mg/dL])
  * Creatinine clearance for females = 0.85 x male value
* Prior treatment with angiotensin receptor blocker (ARB) for hypertension is allowed. If the patient is randomized to a non-losartan containing treatment arm, the patient must be changed to an antihypertensive medication that is not in the class of angiotensin receptor blocker (ARB).
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy within 6 months are eligible for this trial.
* Participants with evidence of chronic hepatitis B virus (HBV) infection on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment are eligible even if they do not have an undetectable HCV viral load.
* Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* The effects of treatment are harmful on the developing human fetus are unknown. For this reason, all patients of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 9 months after completion of mFOLFIRINOX administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Patients with known history of UGT1A1 gene polymorphism detection are eligible to participate. Sites are required to follow the FDA-approved label guidance for Irinotecan when administrating as part of the FOLFIRINOX regimen.

Exclusion Criteria:

* Any prior chemotherapy, radiation therapy, immunotherapy, biologic ('targeted') therapy or investigational therapy for pancreas adenocarcinoma. No prior adjuvant or neoadjuvant therapy for localized pancreatic adenocarcinoma is allowed.
* Patients with deleterious or suspected deleterious germline or somatic BRCA-mutated pancreatic cancer.
* Patients with TRK (tropomyosin receptor kinase) fusion-positive cancers.
* Patients with deficient mismatch/microsatellite unstable or high tumor mutation burden cancers.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* The investigator(s) must state a medical or scientific reason if participants who have brain metastases will be excluded from the study.
* History of allergic reactions attributed to compounds of similar chemical composition to 9-ING-41, losartan, 5-fluorouracil, irinotecan and oxaliplatin not amenable to institutional chemotherapy desensitization protocol. Prior topical fluoropyrimidine use is allowed.
* Patients with cardiac ventricular arrhythmias requiring antiarrhythmic therapy, or atrioventricular heart block (due to 5FU administration)
* Known, existing uncontrolled coagulopathy. Concomitant treatment with full dose warfarin (coumadin) is NOT allowed. Patients may receive low molecular weight heparin (LMWH) (such as enoxaparin and dalteparin) and direct oral anticoagulant (DOAC) for management of deep venous thrombosis (DVT).
* Patients taking strong inhibitors of CYP2C19, CYP3A4, and CYP1A2 or strong inducers of CYP3A4 should only be entered into the study protocol if deemed by the investigator to be in their best interest and with study medical coordinator agreement
* Concomitant use of cimetidine, as it can decrease clearance of 5FU. Another H2-blocker or proton pump inhibitor may be substituted before study entry.
* Participants with uncontrolled intercurrent illness.
* Participants with uncontrolled seizures, central nervous system disorders or psychiatric illness/social situations that would limit compliance with study requirements.
* Known history of active TB (Mycobacterium Tuberculosis).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed. COVID non-live vaccines are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Date of study entry to the earliest date of progressive disease up to 30 months
  Defined from the date of study entry to the earliest date of progressive disease while receiving complete therapy with FOLFIRINOX-based therapy or death due to any cause. PFS will be censored at the date of last follow-up for patients alive without documented progression. PFS curves will be estimated by the Kaplan-Meier method and compared to historical controls treated with FOLFIRINOX alone using the one-sample log-rank test.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 30 months
  Defined from the date of study entry to the date of death due to any cause and censored at the date of last follow-up for patients still alive. OS curves will be estimated by the Kaplan-Meier method and compared to historical controls using the one-sample log-rank test.
Median time of maintenance therapy (mMT): | Up to 30 months
  Defined from the date of starting maintenance 5FU-based therapy to time of objective disease progression.
Objective Response Rate | Up to 30 months
  Defined as the proportion of patients who have a partial or complete response per RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Colin D Weekes, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - University of Washington School of Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Lin EW, Pathak P, O'Shea A, Awasthi B, Phillips IE, Kocher JR, Song Y, Raabe MJ, Xu KH, Patel BK, Lester N, Bae JW, Zhang ML, Nieman LT, Blaszkowsky LS, Walsh EP, Parikh AR, Hansen A, Caufield J, Newbert G, Asombang AW, Casey B, Cohen J, Jacobson BC, Krishnan K, Uppot R, Weissleder R, Horick NK, Hwang WL, Harisinghani MG, Ting DT, Weekes CD. Therapeutic Targeting of Epithelial Mesenchymal Cellular Plasticity in Pancreatic Cancer. Clin Cancer Res. 2025 Dec 9. doi: 10.1158/1078-0432.CCR-25-2052. Online ahead of print. PMID 41364739